CLINICAL TRIAL: NCT06533631
Title: Measuring Brain Health Using Low-Field Portable MRI
Acronym: MR SCREEN
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2000037836; 1R21NS138995-01 (NIH)
Record Dates: First submitted 2024-07-19; First posted 2024-08-01 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: White Matter Hyperintensity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- pMRI and 3T MRI: Participants will receive both a pMRI and high-field 3T MRI at a single study visit for the purpose of comparing WMH measurements against a gold standard (3T MRI).
  Interventions: Device: Portable low-field MRI (pMRI); Device: 3T MRI

INTERVENTIONS:
Device: Portable low-field MRI (pMRI) — Participants will receive a pMRI during the study visit.
Device: 3T MRI — Gold standard MRI for WMH. Participants will receive a 3T MRI during the study visit.

SUMMARY:
The purpose of this study is to develop a new grading scale and utilize automated segmentation for measurement of White Matter Hyperintensity (WMH) volume using a low field MRI.

DETAILED DESCRIPTION:
This study will take place in one visit, if feasible. This visit will take approximately 2 hours. (Alternatively, the visit can be split over two visits if the subject cannot tolerate two consecutive scans. The pMRI and 3T MRI can occur up to one month apart.)

The purpose of this study is to create both a qualitative lowfield WMH scale that can be used widely and a machine learning enabled quantitative measurement of WMH for more sophisticated applications. To ensure the reliability of these WMH measurement systems, participants will receive both a pMRI and high-field 3T MRI at a single study visit for the purpose of comparing WMH measurements against a gold standard (3T MRI). Using the Delphi method, an expert panel of pMRI researchers will develop the low-field WMH grading scale, iteratively refine it, and validate it within this cohort. Parallel to this, advanced machine learning methodologies will be utilized in this cohort, allowing for precise quantification of WMH volume on pMRI.

ELIGIBILITY:
Inclusion Criteria:

* One vascular risk factor, from the following:

  1. Hypertension (defined as taking an antihypertensive medication)
  2. Hyperlipidemia (defined as taking a statin or PCSK9 inhibitor)
  3. Diabetes (defined as taking a medication to prevent hyperglycemia)

Exclusion Criteria:

* 1. History of stroke
* History of dementia or other cognitive impairment
* Pacemaker or other MRI contraindications according to the American College of Radiology guidelines

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants, age 50+, with risk factors for white matter hyperintensities, including hypertension, hyperlipidemia and diabetes. Patients may be identified through flyers distributed among outpatient clinics at Yale-New Haven Hospital for general neurology, internal medicine, and preventive cardiology.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
WMH graded on a low-field WMH scale | 2 hours
  Each pMRI scan will be evaluated by two readers experienced in the adjudication of WMH and the high-field 3T MRI will be adjudicated by a board certified neuroradiologist. WMH will be graded on a low-field WMH scale as minimal, moderate, or severe. The low-field WMH scale will be derived by an expert panel consisting of the study investigators and two more neurologists, a neuroradiologist, and neuropsychologist. Investigators will employ the Delphi method to harness the collective expertise of this panel in developing the novel grading scale.

SECONDARY OUTCOMES:
WMH lesion load (in mm3) | 2 hours
  WMH lesion load will be assessed both global and per white matter region of interest (ROI). These ROIs are defined by FreeSurfer, which maps cortical parcels into corresponding WM segments using geodesic distances. Using the high-field MRI as ground truth, investigators will use two metrics to evaluate the WMH in pMRI. The first, and main validation criterion, is the Spearman correlation coefficient between lesion loads (both global and per ROI) estimated from pMRI (by the neural network) and from high-field MRI (obtained via manual delineation). And second, the Dice score between the predicted WMH mask in pMRI and the corresponding ground truth from the high-field MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Adam H de Havenon, MD, Principal Investigator — Yale University
Locations (1):
- Yale Magnetic Resonance Research Center (MRRC) at The Analyn Center (TAC), New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No